CLINICAL TRIAL: NCT02400944
Title: Determinants of Bladder Cancer Recurrence Study (The DETER Study)
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 15-047
Record Dates: First submitted 2015-03-06; First posted 2015-03-27 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer
Keywords: MSK Tobacco Cessation Program; smoking exposure; 15-047
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and/or urine sample

GROUPS / COHORTS (1):
- patients with bladder cancer
  Interventions: Behavioral: questionnaires; Other: Saliva and/or urine sample

INTERVENTIONS:
Behavioral: questionnaires — The study questionnaires (baseline and 2 follow-ups) will capture information on how modifiable factors, including the patients' smoking habits and body weight, have changed since last contact. RSA will conduct this interview at a time convenient to the patient either during a scheduled clinic visit or by telephone.
Other: Saliva and/or urine sample — Patients will contribute approximately 5 mL of saliva at baseline, and at the time of their follow-up questionnaires. If the patient declines to contribute a saliva specimen, they can contribute approximately 10mL of urine. Urine is routinely collected from bladder cancer patients for clinically-related tests. We will also collect urine from every participant for whom the sample is not depleted by clinical tests at the end of the day. Saliva/urine specimens will be tested for cotinine which is regarded as the gold standard to detect recent smoking exposure and is widely used to identify active smokers in epidemiologic studies.

SUMMARY:
The purpose of this study is to learn how different lifestyle factors, such as cigarette smoking and body weight, change after a diagnosis of bladder cancer, and how they influence who gets a bladder cancer recurrence and who does not.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old AND
* Histologically-confirmed non-muscle invasive bladder cancer (NMIBC)

Exclusion Criteria:

* Patients are ineligible for the study if they have/had:
* Histologically-confirmed NMIBC diagnosed >36 months prior to enrollment
* Cystectomy prior to enrollment
* Any condition, which in the opinion of the primary MSK clinician or investigators precludes their ability to provide informed consent or comply with study procedures
* Non English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinic
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2015-03; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
recurrence | 1 year
  will be defined as the presence of pathologically-confirmed NMIBC lesion >8 weeks after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Helena Furburg-Barnes, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/